CLINICAL TRIAL: NCT03221972
Title: Vitamin D Nutritional Status and Its Related Factors for Chinese Children and Adolescents in 2010-2012
Brief Title: Vitamin D of Chinese Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Lichen Yang (Other Government)
Responsible Party: Sponsor-Investigator, Lichen Yang, National Institute for Nutrition and Health, Centers for Disease Control and Prevention, China
Organization: Centers for Disease Control and Prevention, China (Other Government)
Other Study IDs: 20120212
Record Dates: First submitted 2017-07-12; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Vitamin D Deficiency
Keywords: 25 hydroxyvitamin D; 6-17 years old; vitamin D deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 2 mL of fasting venous blood was collected and centrifuged at 1500×g for 15 minutes within 30 minutes after blood taken. The upper serum was aliquoted and stored in brown vessel at -20℃ in the laboratory where the investigation point was located. All the serum specimens from all the 150 investigation points were transported to our laboratory by cold chain. All the samples were preserved at -70℃ refrigerator before determination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to assess the vitamin D status and analyze risk factors for vitamin D inadequacy of Chinese children and adolescents aged 6-17y.

DETAILED DESCRIPTION:
In this study, we analyzed the vitamin D status of Chinese children and adolescents aged 6-17y, and related risk factors (such as gender, region strata, ambient UVB level at area of residence, season, and outdoor time, etc.). Serum 25 hydroxyvitamin D [25(OH)D] was measured with a radioimmunoassay kit in 15 000 children and adolescent participants in Chinese national nutrition and health survey (CNNHS) 2010-2012. Age, gender, region type, ethnicity, outdoor time, vitamin D supplementation were recorded in unified design questionnaires. Season was recorded by the date of blood taken; location was divided into north and south by China's Qinling mountains and Huaihe river; and ambient ultraviolet B (UVB) radiation level was classified according to the corresponding dose of each participant living area from National Aeronautics and Space Administration data.

ELIGIBILITY:
Inclusion Criteria:

Participanted in China national nutrition and health survey (CNNHS) 2010-2012; Aged 6-17 years; Had blood taken;

Exclusion Criteria: No.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The participants of this study were aged 6-17y selected from the Chinese national nutrition and health survey
Sampling Method: Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
25 hydroxyvitamin D | through study completion, an average of 1 year
  To describe the vitamin D status,ng/mL.

SECONDARY OUTCOMES:
Demographic data | through study completion, an average of 1 year
  age, gender, ethnicity
Environmental data | up to 25 weeks
  season,region type, latitude, ambient ultraviolet B radiation level
Outdoor time | through study completion, an average of 1 year
  outdoor activity time
Vitamin D supplementation | through study completion, an average of 1 year
  frequency of vitamin D supplements taking for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Lichen Yang, Study Director — National Institute for Nutrition and Health, China CDC
Locations (1):
- National Institute for Nutrition and Health, China CDC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The total database of CNHHS 2010-2012 including the database used in our study cannot be made public before the publication of nutrition survey monographs.

REFERENCES:
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Institute of Medicine (US) Committee to Review Dietary Reference Intakes for Vitamin D and Calcium; Ross AC, Taylor CL, Yaktine AL, Del Valle HB, editors. Dietary Reference Intakes for Calcium and Vitamin D. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK56070/ PMID 21796828
- [Background] Golden NH, Abrams SA; Committee on Nutrition. Optimizing bone health in children and adolescents. Pediatrics. 2014 Oct;134(4):e1229-43. doi: 10.1542/peds.2014-2173. PMID 25266429
- [Result] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Result] Turer CB, Lin H, Flores G. Prevalence of vitamin D deficiency among overweight and obese US children. Pediatrics. 2013 Jan;131(1):e152-61. doi: 10.1542/peds.2012-1711. Epub 2012 Dec 24. PMID 23266927
- [Result] Mansbach JM, Ginde AA, Camargo CA Jr. Serum 25-hydroxyvitamin D levels among US children aged 1 to 11 years: do children need more vitamin D? Pediatrics. 2009 Nov;124(5):1404-10. doi: 10.1542/peds.2008-2041. PMID 19951983
- Available data/document: Study Protocol — http://www.chinanutri.cn/gzrw_132/zgjmyyyjkzkjcxm/201412/t20141229_108493.html